CLINICAL TRIAL: NCT00633048
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NSA-789 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating the Safety and Tolerability of NSA-789
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trials Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3230A1-1000
Record Dates: First submitted 2008-02-08; First posted 2008-03-11 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: ascending single-dose study; healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSA-789 (Experimental): active drug
  Interventions: Drug: NSA-789
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NSA-789
  Arms: NSA-789
Drug: placebo
  Arms: placebo

SUMMARY:
This is the first time that NSA-789, a new compound being developed for schizophrenia, will be given to humans. Each healthy subject will receive a single dose, except for 8 subjects who will receive 2 doses-- one dose under fasting conditions and one dose after eating food.

ELIGIBILITY:
Inclusion:

* Healthy men and women between 18 and 50 years old.
* Women must be of non-child-bearing potential (not able to have children).
* Must be of normal body weight.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability from reported adverse events, scheduled physical examinations, vital signs, cardiac rhythm monitoring, 12-lead ECGs, and clinical laboratory test results | 3 months

SECONDARY OUTCOMES:
pharmacokinetics | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tacoma, Washington, United States